CLINICAL TRIAL: NCT05484362
Title: Acute Effect of Two Doses of Crocus Sativus on Postprandial Glycemia: A Randomized Clinical Trial in Healthy Humans
Brief Title: Acute Effect of Crocus Sativus on Postprandial Glycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agricultural University of Athens (Other)
Responsible Party: Principal Investigator, Aimilia Papakonstantinou, Assistant Professor, Agricultural University of Athens
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: HRBD 58/21.06.2022
Record Dates: First submitted 2022-07-30; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Potential Abnormality of Glucose Tolerance; Appetitive Behavior; Blood Pressure
Keywords: Crocus sativus; Blood glucose responses; blood pressure; subjective appetite; blood glucose concentrations
MeSH Terms: conditions — Appetitive Behavior | interventions — Beverages

STUDY DESIGN:
Intervention Model Description: Crossover, double blind, randomized clinical trial
Who Masked: Participant, Investigator
Masking Description: A researcher not involved in data analyses was responsible for participant allocation and test food consumption.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Glucose as reference food (Experimental): Eleven healthy subjects (male: 6, female: 5) after 10-14h fast, consumed 50 g D-glucose, three times, in different weeks along with 250 mL water; and 50 g D-glucose containing 15 mg and 30 mg of Crocus Sativus tested once, in different weeks along with 250 mL water. Fingertip capillary blood glucose samples were taken at 0, 15, 30, 45, 60, 90 and 120 min postmeal. The first glucose sample was taken exactly 15 min after the beginning of the consumption of the tested beverage.
  Interventions: Other: D-Glucose beverage as reference food; Other: 15mg of Crocus Sativus as beverage; Other: 30mg of Crocus Sativus as beverage
- 15mg of Crocus Sativus as beverage (Experimental): Eleven healthy subjects (male: 6, female: 5) after 10-14h fast, consumed 50 g D-glucose, three times, in different weeks along with 250 mL water; and 50 g D-glucose containing 15 mg and 30 mg of Crocus Sativus tested once, in different weeks along with 250 mL water. Fingertip capillary blood glucose samples were taken at 0, 15, 30, 45, 60, 90 and 120 min postmeal. The first glucose sample was taken exactly 15 min after the beginning of the consumption of the tested beverage.
  Interventions: Other: D-Glucose beverage as reference food; Other: 15mg of Crocus Sativus as beverage; Other: 30mg of Crocus Sativus as beverage
- 30mg of Crocus Sativus as beverage (Experimental): Eleven healthy subjects (male: 6, female: 5) after 10-14h fast, consumed 50 g D-glucose, three times, in different weeks along with 250 mL water; and 50 g D-glucose containing 15 mg and 30 mg of Crocus Sativus tested once, in different weeks along with 250 mL water. Fingertip capillary blood glucose samples were taken at 0, 15, 30, 45, 60, 90 and 120 min postmeal. The first glucose sample was taken exactly 15 min after the beginning of the consumption of the tested beverage.
  Interventions: Other: D-Glucose beverage as reference food; Other: 15mg of Crocus Sativus as beverage; Other: 30mg of Crocus Sativus as beverage

INTERVENTIONS:
Other: D-Glucose beverage as reference food — Eleven healthy subjects (male: 6, female: 5) after 10-14h fast, consumed 50 g D-glucose, three times, in different weeks along with 250 mL water; and 50 g D-glucose containing 15 mg and 30 mg of Crocus Sativus tested once, in different weeks along with 250 mL water. Fingertip capillary blood glucose samples were taken at 0, 15, 30, 45, 60, 90 and 120 min postmeal. The first glucose sample was taken exactly 15 min after the beginning of the consumption of the tested beverage.
Other: 15mg of Crocus Sativus as beverage — Eleven healthy subjects (male: 6, female: 5) after 10-14h fast, consumed 50 g D-glucose, three times, in different weeks along with 250 mL water; and 50 g D-glucose containing 15 mg and 30 mg of Crocus Sativus tested once, in different weeks along with 250 mL water. Fingertip capillary blood glucose samples were taken at 0, 15, 30, 45, 60, 90 and 120 min postmeal. The first glucose sample was taken exactly 15 min after the beginning of the consumption of the tested beverage.
Other: 30mg of Crocus Sativus as beverage — Eleven healthy subjects (male: 6, female: 5) after 10-14h fast, consumed 50 g D-glucose, three times, in different weeks along with 250 mL water; and 50 g D-glucose containing 15 mg and 30 mg of Crocus Sativus tested once, in different weeks along with 250 mL water. Fingertip capillary blood glucose samples were taken at 0, 15, 30, 45, 60, 90 and 120 min postmeal. The first glucose sample was taken exactly 15 min after the beginning of the consumption of the tested beverage.

SUMMARY:
This study investigated the effects of two different doses of Crocus Sativus in glucose beverages on glycemic responses.

DETAILED DESCRIPTION:
This study examined the short-term effects of two different doses (15 mg and 30 mg) of Crocus Sativus in glucose beverages on postprandial glycemic responses in healthy young adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non-smoking
* Non-diabetic men and women
* Body Mass Index (BMI) between 18.5 and 24.9 kg/m2
* Normal blood pressure

Exclusion Criteria:

* Severe chronic disease (e.g., coronary heart disease, diabetes mellitus, kidney or liver conditions, endocrine conditions)
* Gastrointestinal disorders
* Pregnancy
* Lactation
* Competitive sports
* Alcohol abuse
* Drug dependency
* Allergy in Crocus Sativus

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Capillary blood glucose responses | 2 hours
  Clinically useful change in blood glucose, defined as the restoration of glucose within normal limits during the 2-hour oral glucose tolerance test

SECONDARY OUTCOMES:
Subjective appetite ratings | 2 hours
  Useful change in subjective appetite using visual analogue scales with a score from 0 to 10 (given in the form of booklet, one scale per page) at baseline, 15, 30, 45, 60, 90 and 120 min. The minimum or maximum score will be evaluated if it is better or worse depending on the appetite variable e.g., hunger, satiety, desire to eat etc.
Blood pressure | 2 hours
  Useful change in systolic and diastolic blood pressure before and 2-hour after consumption of the three beverages

CONTACTS AND LOCATIONS:
Overall Officials: Aimilia Papakonstantinou, PhD, Principal Investigator — Agricultural University of Athens
Locations (1):
- Agricultural University of Athens, Athens, Attica, Greece